CLINICAL TRIAL: NCT05225064
Title: Increasing COVID-19 Vaccine Uptake in Developing Countries (Bihar)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Connecticut (Other); Lahore University of Management Sciences (Other); University of California, Berkeley (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000031541
Record Dates: First submitted 2022-02-02; First posted 2022-02-04 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Vaccination Refusal
Keywords: COVID-19; vaccination; masks; incentives
MeSH Terms: conditions — Vaccination Refusal; COVID-19 | interventions — Masks

STUDY DESIGN:
Intervention Model Description: There are five arms. Arm 1: Control; Arm 2: Village-level vaccine clinics with monetary, non-monetary, or no incentive; Arm 3: Household-level vaccination with monetary, non-monetary, or no incentive; Arm 4: Mask promotion; Arm 5: Village-level vaccine clinics and mask promotion
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will be blind to study arm assignment. Due to the nature of the intervention, participants and care providers will not be blind to intervention assignment; however they are likely to be unaware of intervention components because they are not expect to communicate with those who are assigned to a different intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): No vaccine or mask promotion, but access to vaccines increased to match access in intervention villages
- Village-level vaccine clinics with monetary, non-monetary, or no incentive (Experimental): Village-level vaccine clinics with monetary, non-monetary, or no incentive. Villages are cross-randomized to grocery coupon, food ration, no incentive, or grocery coupon to both community member and community health worker after the community member has received a vaccination.
  Interventions: Behavioral: Incentives to be vaccinated; Behavioral: Vaccination made more convenient; Behavioral: Social mobilization campaign to be vaccinated
- Household-level vaccination with monetary or no incentive (Experimental): Household-level vaccination with monetary incentive or no incentive. Villages are cross-randomized to grocery coupon or no incentive upon receiving vaccination
  Interventions: Behavioral: Incentives to be vaccinated; Behavioral: Vaccination made more convenient; Behavioral: Social mobilization campaign to be vaccinated
- Village-level vaccination without incentive, plus mask promotion (Experimental): Individuals are encourage to attend village-level vaccine clinics but not given any incentive. Mask distribution and reinforcement activities are conducted in villages at a similar time as vaccine promotion.
  Interventions: Device: Mask; Behavioral: Encouragement to wear a mask; Behavioral: Vaccination made more convenient; Behavioral: Social mobilization campaign to be vaccinated
- Village-level vaccination without incentive (Experimental): Individuals are encourage to attend village-level vaccine clinics but not given any incentive.
  Interventions: Behavioral: Vaccination made more convenient; Behavioral: Social mobilization campaign to be vaccinated

INTERVENTIONS:
Behavioral: Incentives to be vaccinated — Individuals will be provided with a guaranteed cash payment, entry into a cash lottery, or guaranteed gift of food if they are vaccinated
  Arms: Household-level vaccination with monetary or no incentive; Village-level vaccine clinics with monetary, non-monetary, or no incentive
Device: Mask — Individuals are given cloth masks
  Arms: Village-level vaccination without incentive, plus mask promotion
Behavioral: Encouragement to wear a mask — Individuals who are not wearing masks over their mouth and nose are stopped in public places and encouraged to wear a mask
  Arms: Village-level vaccination without incentive, plus mask promotion
Behavioral: Vaccination made more convenient — Vaccines are conducted at the household-level rather than the village-level
  Arms: Household-level vaccination with monetary or no incentive; Village-level vaccination without incentive; Village-level vaccination without incentive, plus mask promotion; Village-level vaccine clinics with monetary, non-monetary, or no incentive
Behavioral: Social mobilization campaign to be vaccinated — Village-level social mobilization campaign to be vaccinated
  Arms: Household-level vaccination with monetary or no incentive; Village-level vaccination without incentive; Village-level vaccination without incentive, plus mask promotion; Village-level vaccine clinics with monetary, non-monetary, or no incentive

SUMMARY:
Working with governments in Bihar, India, we will evaluate a number of mechanisms to increase vaccine uptake. These include household vaccination visits instead of community vaccination clinic.monetary and non-monetary incentives, and concurrent mask promotion. This ClinicalTrials entry contains results only for the study in Bihar.

DETAILED DESCRIPTION:
The goal of the study is to identify strategies that best promote and support COVID vaccine uptake in developing countries, we propose to test a range of scalable social and behavioural interventions. This could help policy makers design and employ interventions that are effective. This is especially valuable in resource constrained contexts where funds and institutional resources can be diverted towards interventions that have proven to work.

In Bihar the intervention will be village-level social mobilization involving community promotion, including in-person vaccine reinforcement, and household-level social mobilization. Some treatment villages will receive household- level interventions with varying intensity (different proportion of households will be visited). There will also an accompanying mask distribution campaign during household visits where the importance of mask-wearing as a complement to vaccine use will be explained.

This ClinicalTrials entry contains results only for the study in Bihar.

ELIGIBILITY:
Inclusion Criteria:

* Lives in study village

Exclusion Criteria:

* Does not live in study village

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114512 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Percent of individuals who receive the first, second, or third dose of covid vaccine | up to 4 weeks (endline may vary depending on estimated uptake rates)
  Prevalence of vaccination with difference doses

CONTACTS AND LOCATIONS:
Locations (1):
- Project Concern International, Patna, Bihar, India